CLINICAL TRIAL: NCT03796299
Title: Expression of MCM5 in Urine in Patients With Urothelial Cancers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018
Record Dates: First submitted 2018-12-27; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; biomarker; urothelial cancer; cystoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Patients with bladder cancer
  Interventions: Diagnostic Test: Assessment of expression of MCM5 in the urine (ADX Bladder)
- 2: Patients with upper urinary tract cancer
  Interventions: Diagnostic Test: Assessment of expression of MCM5 in the urine (ADX Bladder)
- 3 (control): Controls
  Interventions: Diagnostic Test: Assessment of expression of MCM5 in the urine (ADX Bladder)

INTERVENTIONS:
Diagnostic Test: Assessment of expression of MCM5 in the urine (ADX Bladder) — Each participant will be asked to urinate in a plastic container. Urine will be centrifuged afterwards, then the expression of MCM5 protein will be examined in cells from urine sediment. For this purpose, it is planned to use the Arquer Diagnostics ADXBLADDER test. It is an enzyme linked immunosorbent assay (ELISA) using two monoclonal antibodies directed against two different epitopes. Both antibodies have high affinity and specificity for the MCM5 antigen.

SUMMARY:
In patients with non-muscle-invasive bladder cancer, the development and introduction to the clinical practice of an adequately accurate biomarker may allow to limit the indications for performing control cystoscopy. Thus, it will reduce the discomfort and stress of patients, the risk of complications of the invasive procedure and probably significantly reduce the costs incurred by healthcare systems.

The aim of the present study is to determine the usefulness of the determination of MCM5 protein expression in the urine of patients with urinary bladder or upper urinary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* written consent to participate in the study,
* ability to void and collect >50ml of urine,
* recurrent bladder cancer confirmed by cystoscopy (group 1) or upper urinary tract tumor confirmed by imaging studies (group 2) or no history of urological/gynecological cancers (controls)

Exclusion Criteria:

* urinary tracy infection,
* nephrolithiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients qualified for surgery due to bladder or upper urinary tract tumors and controls.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Expression of MCM-5 in the urine | Within 48 hours after subject enrollment
  Expression of MCM-5 will be determined in urine sediment by Arquer Diagnostics ADXBLADDER test (ELISA test using two monoclonal antibodies directed against epitopes of high affinity and specificity for the MCM5 antigen).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Dept. of Urology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bialek L, Czerwinska K, Fus L, Krajewski W, Sadowska A, Radziszewski P, Dobruch J, Kryst P, Poletajew S. MCM5 urine expression (ADXBLADDER) is a reliable biomarker of high-risk non- muscle-invasive bladder cancer recurrence: A prospective matched case-control study. Cancer Biomark. 2021;30(2):139-143. doi: 10.3233/CBM-200316. PMID 32924986